CLINICAL TRIAL: NCT07340424
Title: A Prospective, Open-label, Single-arm, Exploratory Clinical Trial to Evaluate the Safety and Tolerability of 225Ac-TR2205 Injection in Patients With Triple-negative Breast Cancer.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xiaorong Sun (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Sun, Director of Nuclear Medicine Department, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR2205-305
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Metastatic Triple-negative Breast Cancer (mTNBC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 225Ac-TR2205 Injection (Experimental)
  Interventions: Drug: 225Ac-TR2205 Injection

INTERVENTIONS:
Drug: 225Ac-TR2205 Injection — Patients will receive 225Ac-TR2205 injection administration at an interval of 8 weeks between each dose.

SUMMARY:
This study is a prospective, single-center, single-arm, open-label research. It evaluates the safety and tolerability of 225Ac-TR2205 in patients with triple-negative breast cancer (TNBC), and assesses its radiation dosimetry and initial efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the study and signing of the informed consent form.
2. Female patients aged 18 years and above.
3. Patients with triple-negative breast cancer who have been diagnosed by histopathology [immune histochemistry estrogen receptor (ER) positive rate < 1% is defined as ER negative expression; progesterone receptor (PR) positive rate < 1% is defined as PR negative; human epidermal growth factor receptor 2 (HER2) expression 0-1+ or HER2 ++ but fluorescence in situ hybridization/colorimetric in situ hybridization (FISH/CISH) negative is defined as HER2 negative expression].
4. Patients with metastatic triple-negative breast cancer who have received at least 2 systemic treatments (at least 1 of which is for metastatic disease).
5. Patients with at least 1 measurable lesion (tumor evaluation according to RECIST 1.1).
6. ECOG performance status assessment of 0-1.
7. Clinical significance of hematological toxicity related to previous treatment must recover to ≤ 2 grade, and non-hematological toxicity ≤ 1 grade (except for hair loss).
8. For patients with reproductive potential: 7 days before the first administration, fertile women must confirm that the urine pregnancy test is negative and agree to use effective contraceptive measures during the use of the study drug and within 6 months after the last administration (such as oral contraceptives, intrauterine devices, restraint of sexual desire or barrier contraception combined with spermicides, etc.).

Exclusion Criteria:

1. Patients who received radiotherapy (except palliative radiotherapy) or chemotherapy, immunotherapy within 3 weeks before treatment, except for bisphosphonates (which can be used for bone metastasis), are excluded.
2. Patients who received radionuclide therapy within 6 months before enrollment, such as strontium-89, samarium-153, rhenium-186, rhenium-188, radium-223, lutetium-177, actinium-225, or whole-body radiotherapy.
3. Patients who are undergoing chemotherapy, immunotherapy, biological therapy, off-label radionuclide therapy, or other investigational treatments.
4. Patients who have undergone major surgery within 28 days before enrollment.
5. Patients evaluated by the investigator are expected to have a life expectancy of less than 3 months.
6. Bone scans show super bone imaging, defined as uniform and significant concentration of radioactive isotopes in the entire skeleton relative to soft tissue, while the urinary system is not visible or shows mild visibility.
7. Symptomatic spinal cord compression, or clinical or imaging evidence suggesting impending spinal cord compression.
8. Patients with uncontrollable central nervous system (CNS) metastases, who need symptomatic treatment with glucocorticoids or mannitol, and if necessary, enhanced CT or MRI to clarify the status of brain metastases.
9. Patients with a history of other malignant tumors, except for those with fully treated malignant tumors that have survived without treatment for more than 3 years without recurrence or progression, or patients with fully treated non-melanoma skin cancer and superficial bladder cancer.
10. Patients with a history that may interfere with the purpose of the study and assessment, or the investigator determines that the patient has any condition that cannot cooperate with imaging examinations, treatment, and procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity grades of adverse events (AE), serious adverse events (SAE), and unexpected serious adverse reactions (SUSAR) were evaluated according to the CTCAE 5.0 standard. | 8 weeks after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China